CLINICAL TRIAL: NCT05452434
Title: Mirabegron Combined With Behavioral Intervention for Overactive Bladder：a Prospective Multicenter Randomized Controlled Clinical Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Honghui Shi, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShiHH
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 300 cases, mirabegron 50mg QD + behavior intervention (timed urination + left head wagging 3 times and right head wagging 3 times in urgent urination) for 12 weeks.
  Interventions: Drug: mirabegron
- Control group (Active Comparator): 300 cases, mirabegron 50mg QD for 12 weeks
  Interventions: Drug: mirabegron

INTERVENTIONS:
Drug: mirabegron — mirabegron 50mg QD for 12 weeks.

SUMMARY:
The purpose of this study was to assess the efficacy, safety and tolerability of Mirabegron and behavioral combination versus Mirabegron alone in the treatment of women with overactive bladder (OAB）.

ELIGIBILITY:
Inclusion Criteria:

* 1. Female aged between 40-60 years old, and no abnormalities were found in general examination, neurological examination and pelvic examination. 2. Patients with urgent urination for more than 3 months, with or without urgent incontinence, often with frequent micturition and nocturia, have normal urine routine. 3. The patients who were diagnosed as OAB by the following questionnaires, with 6≤ score ≤11 is moderate OAB, with score≥12 is severe OAB, and selected moderate and severe OAB patients. 4. Willing to join the study with signed ICF.

Exclusion Criteria:

* 1. Other diseases as obvious reasons causing OAB symptoms. 2. Patients with hypertension, of whom blood pressure is as high as 180/110 mm Hg or above. 3. Patients with gynecological malignancies, pelvic radiation therapy, stress urinary incontinence or mixed urinary incontinence with predominant stress incontinence. 4. Those taking OAB treatment drugs; 5. Pregnant (blood G-HCG determination if necessary) or lactating women; 6. Women with liver and kidney dysfunction, immunosuppressive agents, blood diseases, diabetes, mental illness or other serious diseases. 7. Poor compliance. 8. Allergic constitution, or allergic to the type of study drug

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Overactive Bladder Symptom Score (OABSS) Total Score | From first dose of study drug up to month 9

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first dose of study drug up to month 9